CLINICAL TRIAL: NCT07076108
Title: The Safety and Efficacy of Oral Vitamin C Administration on Erythropoietin Dosing Requirement in End-Stage Renal Disease Patients on Regular Hemodialysis
Brief Title: Oral Vitamin C Administration on Erythropoietin Dosing Requirement in End-Stage Renal Disease Patients on Regular Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, marwa hassan, Faculty of Pharmacy, Ain Shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 252
Record Dates: First submitted 2025-07-13; First posted 2025-07-21 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Vitamin C; Oral Administration; Erythropoietin; End-Stage Renal Disease; Regular Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): Patients were on normal regimen of treatment of anemia.
  Interventions: Drug: Normal regimen of treatment of anemia
- Group B (Experimental): Patients were on 250 mg oral vitamin C daily for 3 months.
  Interventions: Drug: Vitamin C
- Group C (Experimental): Patients were on 500 mg oral vitamin C daily for 3 months.
  Interventions: Drug: Vitamin C

INTERVENTIONS:
Drug: Normal regimen of treatment of anemia — Patients were on normal regimen of treatment of anemia.
  Arms: Group A
Drug: Vitamin C — Patients were on 250 mg oral vitamin C daily for 3 months.
  Other Names: 250 mg oral vitamin C
  Arms: Group B
Drug: Vitamin C — Patients were on 500 mg oral vitamin C daily for 3 months.
  Other Names: 500 mg oral vitamin C
  Arms: Group C

SUMMARY:
The study aimed to evaluate the safety and efficacy of oral vitamin C administration on erythropoietin dosing requirement in end-stage renal disease patients on regular hemodialysis.

DETAILED DESCRIPTION:
Erythropoietin deficiency is the most significant cause of anemia in chronic kidney disease (CKD) and has been demonstrated to occur at each stage of kidney failure. Because the kidney is the sole source of erythropoietin (EPO) synthesis in adults, reduction in kidney mass as occurs in progressive CKD often results in impairment of EPO production, resulting in anemia.

Vitamin C deficiency can interfere with iron absorption and utilization, as well as lead to various abnormalities. The occurrence of widespread vitamin C deficiency in dialysis patients calls for greater attention to these clinical problems. Ascorbic acid is low in patients with advanced CKD and end-stage renal disease (ESRD) due to dietary restrictions on vitamin C-rich foods, as these foods are usually also rich in potassium.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Both sexes.
* Stable hemodialysis (HD) for 90 days or more
* Hemoglobin (HB) levels of 9-11 g/dL (as Hb levels above 11 g/dL, Epo dose reduction is recommended irrespective of iron level).
* Erythropoietin (EPO) dose ≥4000 U/HD session and unchanged dose for two consecutive months
* Ferritin level >100 mcg/L.
* Transferrin saturation (Tsat) of <30 %.
* Not on a vitamin C supplement.
* Not receiving iron supplementation in the preceding 2 months. Each patient's previous 2-month stable dose of Epo was taken as the control.

Exclusion Criteria:

* Patients with gastrointestinal bleeding.
* Blood transfusion, malignancy.
* Hospital admission or history of noncompliance with dialysis and/or medication were excluded from the study and were also censored if these events occurred during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-04-28 (Actual)

PRIMARY OUTCOMES:
Hemoglobin level | 3 months post-procedure
  Hemoglobin level was assessed every month for 3 months

SECONDARY OUTCOMES:
Serum iron level | 3 months post-procedure
  Serum iron level was assessed every month for 3 months
Transferrin saturation | 3 months post-procedure
  Transferrin saturation was assessed every month for 3 months
Change in erythropoietin dose | 3 months post-procedure
  Change in erythropoietin dose was assessed every month for 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.